CLINICAL TRIAL: NCT06675682
Title: Acute Ingestion of Beetroot Juice Does Effects on Contractile or Neuromuscular Properties in Male Trained Sprinters: a Randomized, Double-blind, Placebo-controlled Study.
Brief Title: Beetroot Juice Effects on Contractile or Neuromuscular Properties in Male Trained Sprinters
Acronym: BEET_SPRINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pontificia Comillas (Other)
Collaborators: Universidad Francisco de Vitoria (Other); Universidad de León (Other); Anglia Ruskin University (Other); Universidad Rey Juan Carlos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UPC_Comillas
Record Dates: First submitted 2024-08-27; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-08

CONDITIONS: Nitrates; Placebo
Keywords: Sport nutrition; Track and field; Tensiomyography; Athletes; Nitrates
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beetroot juice supplementation (Experimental): One serving 70 mL of beetroot juice (6.4 mmol of NO3-; Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) 2.5 h before initiating the testing session.
  Interventions: Dietary Supplement: Beetroot Juice (Beet-It Stamina Shot) and Exercise Training
- Placebo supplementation (Placebo Comparator): One serving 70 mL of beetroot juice placebo (0.04 mmol of NO3-; Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) 2.5 h before initiating the testing session.
  Interventions: Dietary Supplement: Beetroot Juice (Beet-It Stamina Shot) and Exercise Training

INTERVENTIONS:
Dietary Supplement: Beetroot Juice (Beet-It Stamina Shot) and Exercise Training — Player randomization was performed using an online tool (https://www.randomizer.org/). An independent researcher assigned alphanumeric codes to each sequence to ensure blinding of both sprint athletes and researchers during the trials. Each player participated in two identical experimental trials separated by one week to allow physical recovery between testing occasions and washout from the beetroot juice treatment.

SUMMARY:
Beetroot juice is a rich source of nitrate (NO3-), which serves as a precursor to nitric oxide (NO) via the NO3- to nitrite (NO2-) to NO conversion pathway. This pathway is believed to enhance vasodilation and improve neuromuscular function, such as by increasing sarcoplasmic reticulum calcium release and re-uptake, leading to enhanced force production in type II muscle fibers and improved muscle contractile recruitment. Therefore, the aim of this study was to investigate the effects of beetroot juice supplementation on muscle contractile properties, as assessed by tensiomyography, and neuromuscular performance in sprint-trained athletes.

DETAILED DESCRIPTION:
Sports nutrition is a rapidly expanding scientific field that has experienced a significant increase in interest from the academic community over the past decade. Despite the extensive marketing of numerous nutritional products that claim to optimize athlete health, function, and performance, only a limited number of sports foods or dietary supplements have been supported by robust evidence for enhancing performance. Among these, caffeine, creatine, beetroot juice, β-alanine, and bicarbonate are notable for their validated efficacy, though the effectiveness of these supplements can vary based on the specific event, context of use, and the individual athlete's goals and responsiveness.

Beetroot juice, in particular, is a rich source of nitrate (NO3-), which serves as a precursor to nitric oxide (NO) through the NO3- to nitrite (NO2-) to NO conversion pathway. This pathway is believed to promote vasodilation and improve neuromuscular function, such as by increasing sarcoplasmic reticulum calcium release and re-uptake, leading to enhanced force output in type II muscle fibers and improved muscle contractile recruitment. Therefore, the aim of this study was to investigate the effects of beetroot juice supplementation on muscle contractile properties, as assessed by tensiomyography, and neuromuscular performance in sprint-trained athletes. The goal was to gain a deeper understanding of the physiological effects induced by beetroot juice intake in short-distance track and field disciplines.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 to 40 years old.
* With a regular training practise in track and field disciplines > 5 years.

Exclusion Criteria:

* Intolerance to beetroot juice or NO3- derivatives
* Presence of any chronic pathology or injury within three months prior to the study-
* Use of medications or supplements (e.g., caffeine) during the study.
* Failure to attend all experimental sessions.
* Failure to adhere to the dietary guidelines established in the study

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Tensiomyography changes (seconds): Delay time (Td) ; Contraction time (Tc) ; Sustain time (Ts) ; Relaxation time (Tr) | 1-week
  The measurement of the rectus femoris, biceps femoris, gastrocnemius lateralis, and gastrocnemius medialis muscles was conducted using tensiomyography. We analyzed different parameters such as selay time (Td) as a time between the electrical impulse and 10% of the contraction; Contraction time (Tc) as a time between 10% and 90% of the contraction; Sustain time (Ts) as a time between 50% of the contraction and 50% of the relaxation; Relaxation time (Tr) as a time between 90% and 50% of the relaxation.
Changes in 60-m and 100-m sprint test (seconds) | 1-week
  Time to complete 60-m and 100-m sprint test using photocell timing gates

SECONDARY OUTCOMES:
Changes in maximal countermovement and squat jump height (cm) | 1-week.
  Maximal jump height using a contact platform
Changes in nitrites and nitrates levels in saliva (μmol/L) | 1-week
  Using specific kit ELISA analysis
Changes in side effects questionnarie | 1-week
  Questionnarie based on side-effects related to beetroot juice ingestion (A scale consisting of nine items, each answered with "yes" or "no")
Changes in rate of perception effort | 1-week
  Using rate of perceived exertion scale (1-10 points)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro López Samanes, PhD, Study Director — Universidad Pontificia Comillas
Locations (1):
- Universidad Pontificia Comillas, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided